CLINICAL TRIAL: NCT04031924
Title: An Evaluation of Balance, Functional Capacity, Kinesiophobia and Physical Fitness in Patients With Liver Transplantation
Brief Title: Kinesiophobia and Physical Fitness, and Related Factors in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Taskin, Clinical physiotherapist, Hacettepe University
Other Study IDs: NACIYEVARDAR
Record Dates: First submitted 2019-07-08; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Liver Transplant Disorder
Keywords: liver transplantation; functional capacity; kinesiophobia; balance; physical fitness; physical activity; muscle strength
MeSH Terms: conditions — Kinesiophobia; Motor Activity | interventions — Physical Fitness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver Transplantation: Sixteen individuals with liver transplantation were included in the study, and their physical and demographic characteristics of the individuals recorded. The Senior Fitness Test (SFT) was used to evaluate to physical fitness. The Tampa Scale for Kinesiophobia (TSK) was used to assess kinesiophobia; the Fatigue Impact Scale (FIS) and Fatigue Severity Scale (FSS) to evaluate fatigue; the Berg Balance Scale (BBS) and the Timed Up and Go test (TUG) to evaluate the balance; the International Physical Activity Questionnaire (IPAQ) to determine the level of physical activity;and the Hospital Anxiety and Depression Scale (HADS) to evaluate psychological status.
  Interventions: Other: Assessment of: 1. Functional Capacity 2. Physical Fitness 3. Physical Activity Level 4. Balance 5. Kinesiophobia 6. Psychological Status 7. Fatigue Severity
- Healthy Subjects: Sixteen age- and sex-matched healthy subjects were included in the study.
  Interventions: Other: Assessment of: 1. Functional Capacity 2. Physical Fitness 3. Physical Activity Level 4. Balance 5. Kinesiophobia 6. Psychological Status 7. Fatigue Severity

INTERVENTIONS:
Other: Assessment of: 1. Functional Capacity 2. Physical Fitness 3. Physical Activity Level 4. Balance 5. Kinesiophobia 6. Psychological Status 7. Fatigue Severity — All liver transplantation patients who underwent transplant at least one year ago and healthy subjects were evaluated the first day they came.

SUMMARY:
Kinesiophobia and Physical Fitness, and Related Factors in Liver Transplantation

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age who had undergone liver transplantation at Hacettepe University Hospital at least one year ago were eligible for the study.

Exclusion Criteria:

* Hepatic encephalopathy
* Progressive cardiac and/or pulmonary disease
* Central nervous system pathologies
* Orthopedic problems preventing physical assessments
* Multiorgan transplantation
* Cognitive deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixteen individuals older than 18 years of age who had undergone liver transplantation at Hacettepe University Hospital at least one year ago and 16 age- and sex-matched healthy subjects were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Physical Fitness | 10 minutes
  The Chair Stand Test: This requires people to repeatedly stand up from and sit down on a chair for 30 seconds. The number of stands is recorded.
Physical Fitness | 10 minutes
  The Biceps Curl Test: This requires people to repeatedly lift a 5 lb(2.27 kg) weight (for women) or an 8 lb (3.63 kg) weight (for men) for 30 seconds. The number of lifts is recorded.
Physical Fitness | 30 minutes
  The 6-minute Walk Test: This is measured in distance (m) and reflects aerobic endurance. The original version of the Senior Fitness Test required people to walk on a straight line.
Physical Fitness | 5 minutes
  The Chair Sit and Reach Test: This is measured in distance (cm) and reflects lower body flexibility.
Physical Fitness | 5 minutes
  The Back Scratch Test: This is measured in distance (cm) and reflects upper body flexibility.
Physical Fitness | 10 minutes
  The 8-Foot Up-and-Go test: This is measured in time (seconds) and reflects agility and dynamic balance.

SECONDARY OUTCOMES:
Kinesiophobia | 15 minutes
  Kinesiophobia was assessed in all participants using the Tampa Scale of Kinesiophobia (TSK). The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
Balance | 20 minutes
  Berg Balance Scale (BBS) was used to evaluate balance. The BBS consists of 14 items which include simple mobility task and that are scored on a scale of 0 to 4. The level of proficiency for each activity, a score of "0" is given if the participant is unable to do the task and a score of "4" is given if the participant can complete the task based on the criterion that has been assigned to it. The maximum total score on the test is 56.
Balance | 15 minutes
  The Timed Up and Go Test was used to assess the balance performance of people during the movement. For the starter position, a participant sits in a chair with standard height, measuring a distance of 3 meters from the chair. The test timer starts by the clinician at the moment the clinician said "go", the participant gets up from a chair, walks 3 meters, turns 180° a designed spot, walks back to the seat, when the participant sits down then the test stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No